CLINICAL TRIAL: NCT00165542
Title: Determination of A-Protein Levels in Adult and Pediatric Brain Tumor Patients
Brief Title: A-protein Levels in Adult and Pediatric Brain Tumor Patients
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mark W. Kieran, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 98-137
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Malignant Childhood Central Nervous System Neoplasm
Keywords: A-protein level; brain tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: A PROTEIN levels in all patients and with all tumor types.
  Interventions: Other: A PROTEIN level

INTERVENTIONS:
Other: A PROTEIN level

SUMMARY:
The purpose of this study is to evaluate the sensitivity and specificity of "A-PROTEIN" levels in patients with brain tumors. A-PROTEIN levels will be analyzed both pre and post treatment. Levels in blood and/or cerebrospinal fluid (CSF) will be analyzed and correlated with the underlying diagnosis and outcome.

DETAILED DESCRIPTION:
* Patients will be identified at the time of presentation to their neurologist, neurosurgeon or oncologist.
* Blood or cerebrospinal fluid will be collected for this study only when they are being collected for other reasons before and after each surgery. Samples will also be collected after any event such as significant change in symptoms or radiographic progression.
* Once the patients condition has been stabilized, samples will be take at regular intervals of >= 1 month. The duration of this study is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients with possible malignant or benign lesions of the central nervous system will be included.
* There are no restrictions with respect to treatment protocols or prior therapy.
* Patients will be identified after presentation to the neurosurgical, neurological or oncologic services at participating centers. Any patient with evidence of a central nervous system tumor will be eligible. Individuals without evidence of CNS tumors are also eligible, in order to provide blinded controls.
* A signed informed consent will be requested and required for participation.
* There is no age, sex, or ethnic origin restrictions in this protocol. Patients who choose not to participate in the study will continue to have their regular care as defined by their treating team. Patients who speak foreign languages are eligible as long a translator can be found to ensure proper consent has been obtained.

Exclusion Criteria: There are no exclusion criteria for this study.

Max Age: 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be identified at the time of presentation to their neurologist, neurosurgeon or oncologist
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 1998-06; Primary Completion 2004-02 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
association between serum A-Protein level class and clinical status | 4 years
  Serum samples were collected when patients were due for clinically indicated phlebotomy. Serum A-PROTEIN levels were determined using a competitive labeled antibody assay and patients were classified into 3 groups: negative <7pM, equivocal 7-9.9 pM and positive >/= 10 pM; Clinical status at the same time of the sample collection was established by MRI scans and patients grouped as either resected/decreased versus stable/increased. The relationship between clinical status and A-PROTEIN level was assessed using general estimating equations. Association was defined as a statistically significant p-value from the regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Mark W Kieran, MD,PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institite, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manley P, Li X, Turner C, Chi S, Zimmerman MA, Chordas C, Gordon A, Baker A, Ullrich NJ, Goumnerova L, Marcus K, Hoffman K, Kieran MW. A prospective, blinded analysis of A-PROTEIN (recoverin or CAR protein) levels in pediatric patients with central nervous system tumors. Pediatr Blood Cancer. 2009 Sep;53(3):343-7. doi: 10.1002/pbc.22017. PMID 19422022